CLINICAL TRIAL: NCT04560491
Title: Intraoperative Examination of Sentinel Node for The Decision of Further Lymphadenectomy in Clinical Early Stage Endometrial Cancer: A Diagnostic Study of Turkish Gynecologic Oncology Group (TRSGO-SLN-003)
Brief Title: Intraoperative Examination of Sentinel Node in Endometrial Cancer (TRSGO-SLN-003)
Acronym: TRSGOSLN003
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, salih taskin, Assoc. Professor, Ankara University
Other Study IDs: TRSGO SLN-003
Record Dates: First submitted 2020-09-18; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Endometrial Cancer; Sentinel Lymph Node
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frozen section: Patients underwent intraoperative sentinel node examination by frozen section
  Interventions: Diagnostic Test: Intraoperative examination of sentinel node
- Scrape cytology: Patients underwent intraoperative sentinel node examination by scrape cytology
  Interventions: Diagnostic Test: Intraoperative examination of sentinel node

INTERVENTIONS:
Diagnostic Test: Intraoperative examination of sentinel node — Intraoperative examination of sentinel node by either frozen section or scrape cytology to detect metastasis and decide for further lymphadenectomy.

SUMMARY:
More than half of the cases with macrometastatic sentinel lymph node (SLN) have non-SLN metastasis and leaving these nodes in-situ may impair the survival. This study assessed the diagnostic accuracy of intraoperative SLN frozen section examination and scrape cytology as a possible solution for management of SLN positive patients. Clinical early stage endometrial cancer patients who underwent SLN algorithm and intraoperative frozen section or scrape cytology to evaluate SLN status for metastasis were analyzed retrospectively. Intraoperative examination findings were compared with final pathology results and diagnostic accuracy of frozen section and scrape cytology were evaluated.

DETAILED DESCRIPTION:
Frozen section: Lymph nodes up to 2 mm were embedded as a whole. Lymph nodes between 2-5 mm were cut in half along their long axis and nodes larger than 5 mm were sliced in neat, parallel slices at 2-3 mm intervals-slicing was perpendicular to the long axis of the node. Then whole of the SLNs were stained with hematoxylin and eosin (H&E) and examined by frozen section.

Scrape Cytology: SLNs were cut into 3-mm-thick pieces along their long axis. If the lymph node was smaller than 3 mm, it was cut in half. Both sides of the pieces were scraped separately by an edge of a glass slide or a lancet gently. Obtained materials were smeared immediately onto a slide and placed in ethanol for fixation. Then, all slides were stained with H&E and examined.

The results were reported to the surgeon as positive (metastatic) or negative with the numbers of lymph nodes. After intraoperative examination, lymph nodes were put into formalin solution and sent for final pathologic examination.

Data analyses were performed using SPSS Version 21.0 (IBM Corporation, Armonk, NYC, USA). Shapiro-Wilk test was performed to determine whether the data were normally distributed. Descriptive statistics of continuous variables were compared between groups using Mann-Whitney U test. The Chi-square test or Fisher's exact test (when chi-square test assumptions do not hold due to low expected cell counts) were used to compare categorical variables between groups. Continuous variables were presented as median and min-max values, whereas categorical variables were presented as number and percentage. A p value of <0.05 was considered statistically significant. Performance of each protocol to predict treatment success was assessed using confidence intervals with respect to sensitivity, specificity, positive predictive value, and negative predictive value.

ELIGIBILITY:
Inclusion Criteria:

* Patients with apparently early stage endometrial cancer whose SLNs were evaluated intraoperatively were included to this study

Exclusion Criteria:

* Patients with gross metastatic disease
* Patients who had contraindications to dyes (iodine allergy or hepatic impairments)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — females older than 18 years old with early stage endometrial cancer
Study Population: Patients with clinical early stage endometrial cancer and underwent sentinel lymph node biopsy with intraoperative examination of sentinel node by either frozen section or scrape cytology.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity for the diagnosis of metastatic lymph node intraoperatively | intraoperative test

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)